CLINICAL TRIAL: NCT00632203
Title: A Randomized Phase 2 Study of Maintenance Temozolomide Versus Observation in Stable or Responding Stage III/IV Non-Small Cell Lung Cancer Patients
Brief Title: Study of Maintenance Temozolomide Versus Observation in Stable or Responding Stage III/IV Non-Small Cell Lung Cancer Patients (Study P05146)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05146
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma, Large Cell; Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma, Large Cell; Carcinoma, Squamous Cell | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temozolomide treatment (Experimental): Subjects will receive temozolomide at a dose of 75 mg/m^2 orally (PO) daily for 21 consecutive days, followed by a 7-day rest period, until progression or up to a maximum of 6 cycles, whichever occurs first.
  Interventions: Drug: Temozolomide
- Observation (No Intervention): Observation

INTERVENTIONS:
Drug: Temozolomide — 5-mg, 20-mg, and 100-mg gel capsules, 75 mg/m^2 PO daily for 21 consecutive days, followed by a 7-day rest period, until progression or up to a maximum of 6 cycles, whichever occurs first.
  Other Names: Temodar®; SCH 52365
  Arms: Temozolomide treatment

SUMMARY:
The main objective of this study is to investigate whether administration of maintenance temozolomide following standard treatment could possibly prevent or delay the onset of brain metastases in patients with controlled non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase 2, open-label, randomized, multicenter study of maintenance temozolomide versus observation in subjects with stable or responding stage III/IV NSCLC to be conducted in conformance with Good Clinical Practices. Subjects will be randomly assigned to a study drug (temozolomide) or observation arm. The study drug will be administered at a dose of 75 mg/m^2 PO daily for 21 consecutive days, followed by a 7-day rest period, until progression or up to a maximum of 6 cycles, whichever occurs first. Subjects completing 6 cycles of treatment will be followed up for incidence of brain metastasis for up to 2 years, or until progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (age >=18 years), of either sex, and of any race.
* Subjects must have stage IV or III with pleural and/or pericardial effusion

histologically confirmed NSCLC.

* Subjects must have completed 2-6 cycles of a standard systemic therapy, with or without radiation therapy, consisting of at least 2 anti-tumor agents as first-line treatment for Stage III/IV disease, and have documented complete response (CR), partial response (PR), or stable disease (SD) per Response Evaluation Criteria in Solid Tumors (RECIST).
* Response must be confirmed within 4-8 weeks of completing first-line chemotherapy. Study treatment must begin within 12 weeks of completing first-line chemotherapy.
* Female subjects of childbearing potential or male subjects with female partner of childbearing potential must agree to use a medically accepted method of contraception or be surgically sterilized prior to Screening, while receiving study drug, and for 30 days after stopping study drug. Female subjects of childbearing potential must have a negative pregnancy test confirmed prior to dosing with study drug.
* Subjects must be free of any clinically relevant disease (other than stage III/IV NSCLC) that would, in the principal investigator and/or Sponsor's opinion, interfere with the conduct of the study or study evaluations.
* Subjects must be able to adhere to the dosing and visit schedules, and agree to report medication taken, concomitant medications, and adverse events (AEs).
* Eastern Cooperative Oncology Group (ECOG) performance status <=2.
* Clinical laboratory tests (complete blood count [CBC], serum chemistries) must be obtained within 14 days prior to randomization and meet specified criteria.

Exclusion Criteria:

* Brain metastases documented on post-chemotherapy magnetic resonance imaging (MRI).
* Documented history of brain metastases.
* Subject has received more than one prior anti-tumor regimen for Stage III/IV disease. "Regimen" refers to single drug or planned combination of two or more anti-tumor therapies. Bevacizumab (Avastin®) as part of a planned sequence of therapy after first-line platinum-containing double regimen is not considered a second regimen. Neo-adjuvant treatment for resectable subjects is not considered a second regimen.
* Subject has used any investigational product within 4 weeks prior to enrollment.
* Subject is currently receiving immunotherapy or chemotherapy, cytotoxic or targeted therapy as treatment for active systemic disease. Bevacizumab (Avastin®) as part of the prescribed standard first-line regimen is allowed.
* Female who is pregnant, or intends to become pregnant, during the study.
* Subject is in a situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Subject is currently participating in any other clinical study, with the exception of observational long-term follow-up.
* Subject is allergic to, or has sensitivity to, the study drug or its excipients.
* Documented symptomatic, progressive or new bone metastases following the first-line chemotherapy with or without radiation therapy (biphosphonate use for prophylaxis or as a maintenance therapy is allowed).
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-03-04 (Actual); Primary Completion 2011-01-06 (Actual); Study Completion 2011-01-07 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Boggs DH, Robins HI, Langer CJ, Traynor AM, Berkowitz MJ, Mehta MP. Strategies to prevent brain metastasis in high-risk non-small-cell lung cancer: lessons learned from a randomized study of maintenance temozolomide versus observation. Clin Lung Cancer. 2014 Nov;15(6):433-40. doi: 10.1016/j.cllc.2014.06.008. Epub 2014 Jun 24. PMID 25069747

RESULTS

PARTICIPANT FLOW:
Groups:
- Temozolomide Treatment: Participants received temozolomide at a dose of 75 mg/m^2 orally (PO) daily for 21 consecutive days, followed by a 7-day rest period per 28-day cycle, until progression or up to a maximum of 6 cycles, whichever occurred first.
Period: Overall Study
Arm/Group | Temozolomide Treatment | Observation
Started | 26 | 27
Completed | 25 | 27
Not Completed | 1 | 0
Not completed — Did not start study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temozolomide Treatment | Observation | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.4) | 65.1 (10.8) | 65.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Brain Metastases
Description: Brain Metastases were defined as radiological evidence of brain metastases on magnetic resonance imaging (MRI).
Time Frame: Up to 12 months (as measured from day 1 of cycle 1 of standard first-line systemic chemotherapy)
Population: Evaluable population, defined as a participant who had at least one post-randomization MRI scan
Measure: Number; unit: participants
Arm/Group | Temozolomide Treatment | Observation
Number analyzed (Participants) | 22 | 23
participants | 4 | 3
Statistical Analysis 1: Comparison: Temozolomide Treatment vs Observation; Test type: Superiority or Other; p = 0.6995, 2-sided Exact Pearson Chi-square Test

2. Secondary Outcome: Time to Radiological Central Nervous System (CNS) Progression
Description: Defined as CNS progression as measured by MRI.
  Time to CNS progression was analyzed using the Kaplan-Meier method.
Time Frame: from Cycle 1 Day 1 of Standard First Line Systemic Therapy to radiological progression or the last known CNS progression-free date
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide Treatment | Observation
Number analyzed (Participants) | 26 | 27
months | NA [14.26 to NA] — NA means "not applicable." The median and upper limit of the confidence interval (CI) could not be calculated because they were not reached before the study termination date. | NA [NA to NA] — NA means "not applicable." The median and CI could not be calculated because they were not reached before the study termination date.

3. Secondary Outcome: Time to Progression
Description: The time to progression (per response evaluation criteria in solid tumors [RECIST]) was analyzed using the Kaplan-Meier method.
  Definitions of response per RECIST:
  Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): A decrease of at least 30% in the sum of the longest
  diameter of target lesions.
  Progressive Disease (PD): An increase of at least 20% in the sum of the longest
  diameter of target lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: from Cycle 1 Day 1 of Standard First Line Systemic Therapy to progression or up to 6 cycles (168 days) of study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide Treatment | Observation
Number analyzed (Participants) | 26 | 27
months | 11.70 [9.03 to 15.80] | 10.68 [8.54 to 12.68]

4. Secondary Outcome: Overall Survival
Description: The overall survival was analyzed using the Kaplan-Meier method.
Time Frame: from Cycle 1 Day 1 of Standard First Line Systemic Therapy to the last time of follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide Treatment | Observation
Number analyzed (Participants) | 26 | 27
months | 27.14 [13.90 to NA] — NA means "not applicable." The upper limit of the confidence interval (CI) could not be calculated because it was not reached before the study termination date. | 22.54 [14.52 to NA] — NA means "not applicable." The upper limit of the CI could not be calculated because it was not reached before the study termination date.

5. Secondary Outcome: Number of Participants With Brain Metastases at First Progression
Description: Brain Metastases were defined as radiological evidence of brain metastases on MRI.
Time Frame: from Cycle 1 Day 1 of Standard First Line Systemic Therapy to the last time of follow-up (up to 6 cycles (168 days) of study treatment)
Population: No analysis was performed due to study termination.
Arm/Group | Temozolomide Treatment | Observation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cancer-related Quality of Life (QoL) as Assessed by The European Organization for Research and Treatment of Cancer (EORTC) QoL Questionnaire C30 Version 3.0 (QLQ-C30), and the EORTC Lung Cancer Module (QLQ-LC13)
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Scores range from 0 -100. For functional and global QoL scales, higher scores mean a better level of function. For symptom-oriented scales, a higher score means more severe symptoms and a decrease in QoL. The EORTC QLQ-LC13 is a 13-item questionnaire developed to supplement the EORTC QLQ-C30 in lung cancer patients. It has a score range 0-100 with higher scores representing an increase in symptoms.
Time Frame: as for outcome 5
Population: No analysis was performed due to study termination.
Arm/Group | Temozolomide Treatment | Observation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Tolerability of Maintenance Temozolomide
Description: Tolerability was defined as number of participants with any adverse event leading to study discontinuation and/or study drug discontinuation.
Time Frame: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Temozolomide Treatment | Observation
Number analyzed (Participants) | 26 | 27
participants | 5 | NA

ADVERSE EVENTS:
Arm/Group | Temozolomide Treatment | Observation
Serious Adverse Events (participants affected / at risk) | 8/26 | 4/27
Other Adverse Events (participants affected / at risk) | 25/26 | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide Treatment (N=26) | Observation (N=27)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
DISEASE PROGRESSION (General disorders) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide Treatment (N=26) | Observation (N=27)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 4 (14) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (9) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 13 (17) | 5 (5)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 0 (0)
VOMITING (Gastrointestinal disorders) | 6 (8) | 2 (2)
ASTHENIA (General disorders) | 2 (2) | 2 (2)
CHEST PAIN (General disorders) | 2 (2) | 3 (3)
CHILLS (General disorders) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 15 (16) | 4 (5)
PAIN (General disorders) | 2 (2) | 1 (2)
PYREXIA (General disorders) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (3) | 1 (1)
SINUSITIS (Infections and infestations) | 4 (5) | 3 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 2 (2) | 0 (0)
WEIGHT DECREASED (Investigations) | 4 (4) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
DIZZINESS (Nervous system disorders) | 5 (5) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2) | 4 (4)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (3) | 3 (3)
DEPRESSION (Psychiatric disorders) | 1 (1) | 5 (5)
INSOMNIA (Psychiatric disorders) | 2 (3) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 7 (7)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (3)

LIMITATIONS AND CAVEATS:
The interpretation of the study results should be taken with caution because of the small sample size due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) agrees not to publish/publicly present any interim results of the study without prior written consent from the Sponsor. The PI further agrees to provide 45 days written notice to the Sponsor prior to

submission, to permit the Sponsor to review copies of abstracts/manuscripts for publication, which report any results of the study. The Sponsor shall have the right to review and comment on any presentation.